CLINICAL TRIAL: NCT07103434
Title: A Feasibility Study on the Efficacy of a VR-based Mindfulness Intervention for Dementia Caregivers in the Home Environment: A Pilot Randomized Control Trial
Brief Title: VR-based Mindfulness for Dementia Caregivers in the Home Environment (Mind-body Interventions)
Acronym: vrmdc
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Lingnan University (Other); Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Qi Wang, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250701
Record Dates: First submitted 2025-07-07; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Dementia; Caregiver Burden of People With Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Due to the nature of this trial, neither the staff, participants nor care provider can be masked to allocation. The data analyst will be blinded after study completion by having the intervention group information coded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR Mindfulness intervention (Experimental): Participants in this arm will have the VR-based MBI app developed by the research team and use wearing the JAPAN JTSK 6th generation upgraded version of 3D virtual reality glasses.
  During briefing session, participants will engage in a 5-10 minute exercise within the VR environment, giving participants the opportunity to explore different natural sceneries provided in the app. This exercise aims to acclimate participants to the VR technology and allow them to select environments for their mindfulness practice at home.
  Participants will be provided with the VR glasses to take home and practice mindfulness for approximately 10-15 minutes daily over the next eight weeks. The app will record their practice time for further analysis.
  Interventions: Behavioral: VR Mindfulness intervention
- Audio-based MBI (Experimental): Participants in the audio-based group attend a briefing session where they will receive information on mindfulness practice.
  Participants will listen to the same 10-15 minute audio-based MBI instruction as provided in the VR-based MBI app everyday for the next eight weeks. The instructions in the audio will be the same as the instructions in the VR-based mindfulness app.
  The only difference between the VR-based MBI and audio-based MBI groups will be the absence of VR technology in the audio-based group.
  Interventions: Behavioral: Audio-based MBI
- Usual Care (Waitlist control) (Other): The third group will be the waitlist control group, who will not attend any briefing session or engage in mindfulness-based interventions during the pilot period. Instead, they will have the opportunity to participate in activities provided by community service centres. The researcher will provide the VR-based MBI to the waitlist control group after they have completed the control period.
  Interventions: Behavioral: Waitlist control

INTERVENTIONS:
Behavioral: VR Mindfulness intervention — Parallel randomized controlled trial
  Arms: VR Mindfulness intervention
Behavioral: Audio-based MBI — Parallel randomized controlled trial
  Arms: Audio-based MBI
Behavioral: Waitlist control — Parallel randomized controlled trial
  Arms: Usual Care (Waitlist control)

SUMMARY:
To explore the feasibility, acceptability, and potential effectiveness among dementia caregivers of the mindfulness-based interventions delivered by VR technology (VR-based MBI) in improving psychological well-being and caregiver-recipient relationship.

This study hypothesized that caregivers in the VR-based MBI group will have a greater improvement in psychological wellbeing than those in the audio-based MBI group and the waitlist care-as-usual group.

This is a 3-arm, parallel, single-blinded, pilot randomised control trial comparing VR-based MBI with audio-based MBI and care-as-usual. The target sample includes 90 caregivers of community-dwelling persons with dementia. Each arm (n=30) will receive an eight-week exercise with instruction, with outcome assessment at baseline, post-treatment,

and 2-month follow-up. Qualitative interviews will also be conducted to assess the feasibility and acceptance. The VR-based MBI group will engage in mindfulness exercises using a mobile app and VR technology, incorporating different natural environments. The intervention duration is eight weeks. The primary outcome is the caregivers' psychological well-being regarding depression, anxiety, and stress. The secondary outcomes include caregiver burden, mindfulness level, quality of life and caregiver-recipient relationship.

Following intention-to-treat analysis, quantitative data on effectiveness will be analysed using between-group t-tests and group-by-time effect size (Cohen's d). The six-step thematic analysis will be utilized for qualitative data. The intervention group will accept the VR-based MBI, rate the intervention as feasible and show significant improvements in outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Primary informal caregivers who spend over four hours/day taking care of a community-dwelling person who has been clinically diagnosed with any type of mild-to-moderate dementia at least 6 months;
* Self-reported psychological distress
* Able to speak and read Cantonese.

Exclusion Criteria:

Have practiced mindfulness-based intervention for at least 3 months in the past;

* Have hearing or visual impairment that cannot practice mindfulness via wearing VR
* glasses embedded in a mobile phone app;

  --Do not own a smart phone that can install the VR-based MBI app;
* Caring for a person with dementia living in a residential care setting;
* Caring a person with severe level of dementia;
* Have been diagnosed with any mental disorder or on-site of psychotic disorders;
* Receiving any other type of mental health intervention;
* Participants with a history of motion sickness (due to the risk of VR triggering motion sickness)
* Unable to understand Cantonese.

sickness)

-Unable to understand Cantonese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression, Anxiety, Stress scale | Baseline (pre-test), immediately post-test, and 2 months post-test
  The Depression, Anxiety, Stress Scale-21 (DASS-21) is a widely used self-report questionnaire designed to assess the negative emotional states of depression, anxiety, and stress. The scale contains 21 items, with seven items allocated to each of the three subscales: Depression, Anxiety, and Stress. Respondents are asked to rate the extent to which they have experienced each symptom over the past week using a 4-point Likert scale, ranging from 0 ("Did not apply to me at all") to 3 ("Applied to me very much, or most of the time"). Higher scores indicate greater levels of emotional distress in the respective domains. The DASS-21 is a shortened version of the original 42-item scale and has demonstrated good reliability and validity across diverse populations. It is commonly used in both clinical and research settings to screen for and monitor changes in symptoms related to depression, anxiety, and stress.
The Chinese Version of the Personal Well-being (ONS4) | Baseline (pre-test), immediately post-test, and 2 months post-test
  The Personal Well-being (ONS4) scale, originally developed by the UK Office for National Statistics (ONS), is a brief self-report measure used to assess subjective well-being across four core domains: life satisfaction, sense of worthwhileness, happiness, and anxiety. Each item is rated on a scale from 0 to 10, with higher scores reflecting greater well-being (except for anxiety, where higher scores indicate greater anxiety). The Chinese version of the ONS4 has been adapted and validated to ensure cultural relevance and linguistic accuracy for use among Chinese-speaking populations. This version maintains the original structure and scoring, allowing for reliable assessment of personal well-being in Chinese contexts. It is widely used in surveys and research to monitor overall well-being and mental health.

SECONDARY OUTCOMES:
Cantonese Zarit Burden Scale Short Version | Baseline (pre-test), immediately post-test, and 2 months post-test
  The Zarit Burden Interview (ZBI) is a widely used self-report instrument designed to assess the level of burden experienced by caregivers of individuals with chronic illnesses or disabilities. The short version of the ZBI consists of 12 items, each rated on a 5-point Likert scale ranging from 0 ("Never") to 4 ("Nearly Always"), with higher scores indicating greater caregiver burden.
  The Cantonese version of the ZBI Short Version has been translated and culturally adapted to ensure its suitability for Cantonese-speaking populations. Validation studies have demonstrated that the Cantonese ZBI Short Version retains strong psychometric properties, including reliability and validity, comparable to the original version. This scale is commonly used in both clinical and research settings in Hong Kong and other Cantonese-speaking regions to evaluate caregiver stress and the impact of caregiving responsibilities.
EuroQol 5-Dimension 5-Level | Baseline (pre-test), immediately post-test, and 2 months post-test
  The EUROHIS-QOL 5-Item Index is a brief, self-report measure designed to assess overall quality of life. Developed from the World Health Organization's Quality of Life instruments (WHOQOL), the EUROHIS-QOL consists of five items that capture core domains of quality of life: general quality of life, general health, energy, daily activities, and personal relationships. Respondents rate each item on a 5-point Likert scale, with higher scores indicating better quality of life. The EQ-5D-5L index scores range from -0.59 to 1, with 1 representing the best possible health state. The index is suitable for use in general populations as well as clinical and research contexts. It has been validated across various languages and cultures, demonstrating good reliability and construct validity as a concise tool for assessing quality of life.
five-facet mindfulness questionnaire | Baseline (pre-test), immediately post-test, and 2 months post-test
  The Five Facet Mindfulness Questionnaire (FFMQ) is a widely used self-report instrument designed to assess individual differences in mindfulness. Developed by Baer et al. (2006), the FFMQ consists of 39 items that measure five distinct facets of mindfulness: (1) Observing (noticing or attending to internal and external experiences), (2) Describing (labeling internal experiences with words), (3) Acting with Awareness (attending to one's activities in the moment), (4) Nonjudging of Inner Experience (taking a non-evaluative stance toward thoughts and feelings), and (5) Nonreactivity to Inner Experience (allowing thoughts and feelings to come and go without getting caught up in them). Each item is rated on a 5-point Likert scale ranging from 1 ("Never or very rarely true") to 5 ("Very often or always true"). Higher scores indicate a greater degree of mindfulness in the respective facet. The FFMQ has demonstrated good reliability and validity across diverse populations and is commonly used
Relationship Closeness Scale | Baseline (pre-test), immediately post-test, and 2 months post-test
  The Relationship Closeness Scale (RCS) is a self-report instrument designed to assess the perceived closeness and interconnectedness between individuals in a relationship, such as romantic partners, friends, or family members. The scale typically consists of several items that measure aspects of emotional closeness, frequency of interaction, and the extent to which individuals influence each other's activities and decisions. Respondents rate each item on a Likert-type scale (e.g., from 1 = "Not at all true" to 7 = "Very true"), with higher scores indicating greater perceived closeness within the relationship. The RCS has demonstrated good reliability and validity in both research and applied settings and is often used to examine the quality and depth of interpersonal relationships.